CLINICAL TRIAL: NCT05237128
Title: Comparing Two Dietary Approaches for Type 2 Diabetes: The LEGEND (Lifestyle Education About Nutrition for Diabetes) Study
Brief Title: The Lifestyle Education About Nutrition for Diabetes (Legend) Study
Acronym: LEGEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00202808; R01DK126898-01A1 (NIH)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
Keywords: Very low-carbohydrate diet; Moderate-carbohydrate plate-method diet; Nutrition therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment and data analysis will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very low-carbohydrate diet (Experimental)
  Interventions: Behavioral: Very low-carbohydrate diet
- Moderate-carbohydrate plate-method diet (Experimental)
  Interventions: Behavioral: Moderate-carbohydrate plate-method diet

INTERVENTIONS:
Behavioral: Very low-carbohydrate diet — Participants in this arm will be taught to manage their type 2 diabetes using a very low-carbohydrate diet, also called a ketogenic or "keto" diet. This diet involves eating non-starchy vegetables, leafy greens, cheese, meats, berries, nuts, and seeds and avoiding starchy foods like pasta, bread, rice, beans, many fruits, etc.
  There will be a core phase and a maintenance phase of this study; the core phase will last for about 4 months and will involve weekly or every other week classes, home assignments, and brief check-in surveys. The maintenance phase will last for the remaining time, with classes and check-in surveys approximately once a month.
  Arms: Very low-carbohydrate diet
Behavioral: Moderate-carbohydrate plate-method diet — Participants in this arm will be taught to manage their type 2 diabetes using a plate-method approach. This diet involves eating different categories of foods based on the proportions of a plate, balancing proteins, vegetables, fruits, starches, and fats.
  There will be a core phase and a maintenance phase of this study; the core phase will last for about 4 months and will involve weekly or every other week classes, home assignments, and brief check-in surveys. The maintenance phase will last for the remaining time, with classes and check-in surveys approximately once a month.
  Arms: Moderate-carbohydrate plate-method diet

SUMMARY:
This study is being completed to compare two dietary approaches for participants with type 2 diabetes. This research will test whether a very low-carbohydrate or a plate-method diet better improves outcomes for blood glucose control and body composition for patients with type 2 diabetes that follow one of these approaches for 12 months.

Participants that meet screening and eligibility will be randomized to one of the two diets. In addition to the diet, study specific visits and assessments will be performed at various timepoints.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes, with current HbA1c > 6.5% and < 12% (self-reported and then measured at screening)
* ability to speak English (this is a group-based intervention)
* ability to engage in light physical activity
* willingness to be randomized to either type of diet

Exclusion Criteria:

* unable to provide informed consent
* substance abuse, mental health, cognitive, or medical condition that would, in the opinion of the investigators, make it difficult for the individual to take part in the intervention, may alter key outcomes, or may require important diet modifications and includes conditions such as hypercalcemia or thyroid dysfunction
* pregnant or planning to become pregnant in the next 12 months, or currently breastfeeding (pregnancy and breastfeeding require modifications to the intervention's dietary approaches)
* current use of weight loss medications (this is likely to alter weight outcomes and may alter other measures)
* history of weight loss (bariatric) surgery or plans for bariatric surgery in the next year
* currently enrolled in a weight loss program or have unalterable plans to enroll in one of these programs in the next year
* vegan or vegetarian
* unwilling or unable to participate in study measurements and group classes
* current use of systemic steroids (self-reported in screening survey; oral or IV systemic steroids excluded. Injected steroids may be permitted depending on frequency and timing of injections with regard to lab assessments (minimum of 2 weeks between injection and blood tests))
* weight above 400 pounds (weight limit for dual-energy X-ray absorptiometry (DEXA) scans)
* history of multiple or recent (within the last four years) kidney stones
* currently following a very low-carbohydrate diet
* unwilling to stop an SGLT2 inhibitor medication if the participant were to be randomized to the very low-carbohydrate diet

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 0 to 12 months
  HbA1c will be measured by standard immunoturbidimetric assay methods and quality control measures at a Clinical Laboratory Improvement Amendments (CLIA) certified lab.

SECONDARY OUTCOMES:
Change in Inflammation based on high sensitivity C-reactive protein (hsCRP) | 0 to 12 months
  High-sensitivity C-reactive protein will be measured with nephelometric methods utilizing latex particles coated with CRP monoclonal antibodies and standardized against a CRP reference preparation.
Change in small particle low-density lipoproteins (LDL) | 0 to 12 months
Change in high-density lipoproteins (HDL) | 0 to 12 months
Change in triglycerides | 0 to 12 months
Change in percent body weight loss | 0 to 12 months
Change in percent body fat on DEXA | 0 to 12 months
  This will be measured by dual-energy X-ray absorptiometry scan
Change in percent lean body mass on DEXA | 0 to 12 months
  This will be measured by dual-energy X-ray absorptiometry scan
Change in bone mineral density in total hip | 0 to 12 months
  This will be measured by dual-energy X-ray absorptiometry scan
Change in bone mineral density in lumbar spine | 0 to 12 months
  This will be measured by dual-energy X-ray absorptiometry scan
Change in serum procollagen type I N propeptide (s-PINP) | 0 to 12 months
Change in serum c-terminal telopeptide of type 1 collagen (s-CTX) | 0 to 12 months
Reduction in diabetes medications using medication effect score (MES) | 0 to 12 months
  The medication effect score is a means of assessing the overall intensity of a patient's diabetes pharmacotherapy based on potency and dosages of medications (Alexopoulos et al., 2021).
Change in HbA1c | 0 to 4 months
  HbA1c will be measured by standard immunoturbidimetric assay methods and quality control measures at a Clinical Laboratory Improvement Amendments (CLIA) certified lab.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Saslow, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - The University of California San Francisco (UCSF), San Francisco, California
  - University of MIchigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saslow LR, Eslamian A, Moran P, Hartogensis W, Mason AE, Kim S, Bauer DC, Griauzde DH, Goldman V, Liu V, Stephens P, Raymond K, Yeung G, Leung C, Hecht FM. Protocol for a randomized controlled trial comparing a very low-carbohydrate diet or moderate-carbohydrate plate-method diet for type 2 diabetes: the LEGEND (Lifestyle Education about Nutrition for Diabetes) trial. Trials. 2023 Jul 20;24(1):463. doi: 10.1186/s13063-023-07512-9. PMID 37475033

DOCUMENTS (1):
  • Informed Consent Form (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT05237128/ICF_000.pdf